CLINICAL TRIAL: NCT00749762
Title: Pulmonary Function During Prone and Supine Positioning in Neonatal Intensive Care Unit (NICU) Infants Requiring Assisted Ventilation
Brief Title: Pulmonary Function During Prone and Supine Positioning in NICU Infants Requiring Assisted Ventilation
Status: Withdrawn | Type: Observational
Why Stopped: Computers/hardware for data collection/storage are outdated and unserviceable.
Sponsor: University of Utah (Other)
Responsible Party: Donald Null M.D., University of Utah / Primary Childrens Medical Center
Other Study IDs: 10831
Record Dates: First submitted 2008-09-08; First posted 2008-09-09 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2010-05

CONDITIONS: Pulmonary Function
Keywords: DURING; PRONE; SUPINE; POSITIONING
MeSH Terms: conditions — Deception

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study seeks to determine in Neonatal Intensive Care Unit (NICU) patients specific improvements in pulmonary function which may occur when an infant is ventilated in the prone as compared to the supine position. Modest improvement in oxygen has been reported to occur with prone positioning, but the exact etiology for this change is not clear. A special incubator designed as an integrated care system allows routine care and the measurement of both patient and ventilator breaths during mechanical ventilation. This study will utilize this device to evaluate in NICU ventilated patients whether specific changes in pulmonary function accompany position changes, and whether these are correlated to a change in pulmonary gas exchange.

DETAILED DESCRIPTION:
Healthy Newborns Pulmonary function and body positioning have been studied in term infants with special attention towards predisposing factors for sudden infant death syndrome.

No difference was seen between prone and supine positioning in functional residual capacity or in effective pulmonary blood flow in 12 normal newborn infants. In 39 healthy newborns, crying vital capacity and peak expiratory flow rate were decreased in prone position, suggesting that in the prone position lung volume is decreased and airway resistance is increased. In another study of 14 infants, prone position resulted in a 5 point (%) higher SpO2 and a 1.5 mL/kg increase in tidal volume, but no change in minute ventilation. In these infants fed while prone, sucking pressure and frequency were increased and suck duration was decreased. Diaphragm thickness appeared to be increased in the prone compared to the supine position, both at end inspiration and end expiration, in 16 healthy term infants undergoing ultrasonography, though SpO2, heart rate and respiratory rate were not different. In a study of an intubated one day old term infant with normal lungs, a novel technique using electrical impedance tomography measured a ventral shift in lung aeration in the prone position, and a dorsal shift in aeration in the supine position.

Healthy Preterm Infants In convalescing healthy premature infants, prone compared to supine positioning has been studied with attention to a possible relationship to the frequency and severity of central apnea (apnea of prematurity).

In one study of 22 preterm infants (mean birth weight and GA: 870 g, 27 wks) with symptomatic apnea and bradycardia, no differences in the frequency of apnea, bradycardia or desaturation episodes were noted between being positioned either prone or supine. However, a previous study in 14 stable preterm infants (mean GA 34 wks) with clinical apnea found an increase in apnea density and periodic breathing in the supine position. Similarly, in 55 infants with birth weight <1kg still on supplemental oxygen, the prone position was associated with a 2 point (%) increase in SpO2 and a decreased frequency of desaturation episodes. Another study saw a 7 mmHg increase in transcutaneous oxygen (TcPO2) associated with prone positioning and a significant decrease in the amount of chest wall asynchrony. Thoracoabdominal synchrony improved in the prone position in a study of 24 preterm infants (mean birth weight and GA: 1020 g, 28wks). One study of 11 infants (mean birth weight and GA: 1525 g, 32 wks) saw no differences in pulmonary function (tidal volume, minute ventilation, pulmonary resistance, dynamic compliance) between prone and supine position. Lung compliance, tidal volume and minute ventilation were higher in the prone position for 10 preterm infants (mean birth weight and GA: 2220 g, 35 wks), but so was total work of breathing. However, two other studies (N=45, N=7) have noted decreased work of breathing associated with the prone position in recovering preterm infants. Of interest, during apnea, the decrease in mean cerebral hemoglobin concentration and mean cerebral blood volume is less when premature infants are in the prone versus supine position.

Preterm Infants on Ventilators In a 1979 study of 14 preterm infants with RDS (mean birth weight and GA: 2250 g, 35 wks) at age 5d, prone compared to supine positioning resulted in a 11 mmHg increase in PaO2, a 50% increase in dynamic lung compliance, and a 22% increase in tidal volume. These improvements were enhanced if the dependent abdomen was unrestricted by suspending the infant in a specialized sling. As part of a study on episodic desaturation, it was noted that at 4 wks post natal age, the frequency of hypoxemic episodes decreased from 1.7 to 0.3 episodes per hour when 6 intubated VLBW infants were studied in the prone versus the supine position (mean birth weight & GA: 810g, 26 wks). This was associated with a 3 point (%) higher baseline SpO2 and a 50% increase in minute ventilation. Desaturation episodes coincided with the onset of infant movement, and prone positioned infants initiated movement less frequently. A larger study of 25 intubated premature infants (mean birth weight and GA: 1633 g, 34 wks) found a 6 mmHg increase in PaO2 when infants were cared for in the prone compared to the supine position. Inspiratory and total pulmonary resistance in prone position were noted to be decreased for mechanical but not for spontaneous breaths in a study of 33 intubated premature infants (median birth weight & GA: 82- g, 27 wks) after 2 weeks of age. A 2 point (%) increase in SpO2 was also noted. Twenty-eight intubated preterm infants (mean birth weight and GA: 1378 g, 30 wks) were studied prone and supine at 38h of age and were found to have lower motor activity scale scores, a 1 point (%) higher SpO2, and, in the 14 infants that experienced desaturation, fewer desaturation episodes in the prone position.

Summary

* Prone positioning appears to decrease movement activity in intubated and non-intubated premature infants and thus decrease the frequency of movement associated desaturation episodes.
* There is modest improvement in oxygenation (SpO2 or PaO2) when positioned prone in intubated and non-intubated premature infants.
* Only 4 published studies could be found (2 study with intubated preterm infants, 2 with non-intubated preterm infants) which examined pulmonary function testing during prone and supine positioning. Three studies reported improvement in pulmonary function with prone position, one study saw no change. The two studies involving intubated premature infants did not demonstrate improvements in the same pulmonary function parameters.

ELIGIBILITY:
Inclusion Criteria:

* Any NICU patient who does not have a major congenital anomaly and is on assisted mechanical ventilation will be eligible for this study.

Exclusion Criteria:

* Healthy patients

Ages: 24 Hours to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: For stable NICU infants who require assisted mechanical ventilation beginning after the 1st 24 hours of life and repeating every 2 to 7 days
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2002-10; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald .Null, M.D., Principal Investigator — University of Utah
Locations (1):
- University of Utah / Primary Childrens Medical Center, Salt Lake City, Utah, United States